CLINICAL TRIAL: NCT06866132
Title: Form, Fit and Function Feasibility Study
Brief Title: Response to an Investigational Device in Patients With Restless Legs Syndrome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Noctrix Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-07
Record Dates: First submitted 2025-03-03; First posted 2025-03-10 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Investigational Device Protocol (Experimental): Participants will use the investigational noninvasive neuromodulation device as instructed over a period of 8 weeks (weeks 3 through 10).
  Interventions: Device: Investigational Noninvasive Neuromodulation Device

INTERVENTIONS:
Device: Investigational Noninvasive Neuromodulation Device — The investigational noninvasive neuromodulation device will be setup by the patient at bedtime and will be used every night. The IRB has established that the investigational device is non-significant risk.

SUMMARY:
This study assesses the tolerability, safety, and impact of an investigational medical device on restless legs syndrome symptoms.

The IRB has established that the investigational device is non-significant risk.

DETAILED DESCRIPTION:
In this 12-week study, participants complete a 2-week baseline (no intervention) followed by 8-weeks of investigational medical device intervention (weeks 3-10) followed by 2-weeks with no intervention (weeks 11-12).

ELIGIBILITY:
Inclusion Criteria:

1. - Subject has signed a valid, IRB-approved informed consent form, can understand the requirements of the study and instructions for device usage, and can converse in English
2. - Subject has received a medical diagnosis of primary restless legs syndrome.
3. - Subject agrees to not change dosage or schedule of any medications that are known to impact RLS symptoms during the study, including RLS medications, antidepressants, sleep medications, or sedative antihistamines.
4. - Subject has moderate-severe RLS symptoms as defined by a score of 15 or greater points on IRLS (International Restless Legs Syndrome Study Group Rating Scale) over the week prior to study entry.
5. - Subject reports that RLS symptoms caused awakenings or interfered with falling back asleep at least 3 nights per week during the month prior to study entry,
6. - Subject reports that RLS symptoms are most significant in lower legs and/or feet.

Exclusion Criteria:

1. - The subject has an active medical device implant anywhere in the body (including but not limited to pacemakers, spinal cord stimulators, deep brain stimulators).
2. - The subject has a metal implant at the site of the study device electrode application (not including knee replacements).
3. - The subject has been diagnosed with epilepsy or other seizure disorder.
4. - The subject has a moderate or severe cognitive disorder or mental illness that would affect his or her ability to participate in the study.
5. - The subject has a known allergy to device materials, electrode gel, polyurethane foam, or lycra (or a severe previous reaction to medical adhesives or bandages).
6. - Subject has any of the following at or near the location of device application: Acute injury, Cellulitis, Open sores
7. - The subject is unable or unwilling to comply with study requirements.
8. - The subject has a medical condition not listed above that may put them at risk.
9. - Subject has prior experience with any neurostimulation devices developed by the study sponsor
10. - Subject has a primary sleep disorder other than RLS that significantly interferes with sleep at the present time (e.g. obstructive sleep apnea stably controlled via CPAP would not be an exclusion).
11. - On nights with no RLS symptoms (if any), subject reports typical sleep onset latency of >60min.
12. - Subject has severe peripheral neuropathy affecting the lower legs and/or subject has neuropathy and is unable to clearly distinguish between symptoms of neuropathy and symptoms of RLS.
13. - Subject reports that bedtime is typically outside of 9pm-3am or reports that bedtime regularly varies by more than 4 hours, such as due to shift work.
14. - During initial device set-up, device does not properly fit the subject or calibrated intensity settings are outside of operational range

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Mean Change in IRLS Rating Scale Score | 10 weeks
  International Restless Legs Syndrome Study Group (IRLS) Rating Scale Score is a participant-rated questionnaire that rates RLS severity from 0-40, where 40 is the most severe. The mean change is assessed from study entry to Week 10.

SECONDARY OUTCOMES:
Mean change in the number of nights with RLS per week | 10 weeks
  This outcome measures the change in subject-reported number of nights with RLS, which ranges from 0 to 7 for each time point assessed. The mean change is assessed from study entry to Week 10. A greater decrease represents a better outcome.
Mean Change in MOS-II | 10 weeks
  The Medical Outcomes Study Sleep Problems Index II (MOS-II) score is a subscale of the participant-rated MOS questionnaire that measures subjective sleep quality. The MOS-I (6-items) and MOS-II (9-items) are the two validated subscales of the 12-item MOS Sleep Scale. Both are scored from 0 to 100, where 100 corresponds to the worst possible sleep problems and 0 corresponds to no sleep problems. The mean change is assessed from study entry to Week 10.
Mean Change in MOS-I | 10 weeks
  The Medical Outcomes Study Sleep Problems Index II (MOS-II) score is a subscale of the participant-rated MOS questionnaire that measures subjective sleep quality. The MOS-I (6-items) and MOS-II (9-items) are the two validated subscales of the 12-item MOS Sleep Scale. Both are scored from 0 to 100, where 100 corresponds to the worst possible sleep problems and 0 corresponds to no sleep problems. The mean change is assessed from study entry to Week 10.
Mean PGI-I score | 10 weeks
  The Patient Global Impressions of Improvement (PGI-I) score assesses the patient's perception of their condition's improvement from study entry, with scores ranging from: Very Much Improved (1), Much Improved (2), Minimally Improved (3), No Change (4), Minimally Worse (5), Much Worse (6), Very Much Worse (7). The mean is assessed at Week 10 relative to study entry.
Percent of Patients Reporting Much Improved or Very Much Improved | 10 weeks
  The Responder Rate is the percentage of subjects with a Patient Global Impressions of Improvement (PGI-I) rating of Much Improved or Very Much Improved relative to study entry. The scores for the Patient Global Impressions of Improvement (PGI-I) are: Very Much Improved (1), Much Improved (2), Minimally Improved (3), No Change (4), Minimally Worse (5), Much Worse (6), Very Much Worse (7).
  This endpoint assesses the responder rate at Week 10.
Mean Change in Periodic Limb Movement Index (PLMI) | 10 weeks
  Mean change in the total number of periodic limb movements (PLMs) per hour of sleep from Weeks 1-2 to Weeks 9-10. A greater decrease in PLMs per hour corresponds to a better outcome.
Mean Change in Sleep Efficiency Percentage | 10 weeks
  Sleep efficiency (SE) is the percentage of the time a person spends asleep relative to the total time dedicated to sleep. A better outcome corresponds to a percentage closer to 100%. This endpoint measures the mean change from Weeks 1-2 to Weeks 9-10.
Mean Change in Minutes Awake after Sleep Onset (WASO) | 10 weeks
  Minutes Awake after Sleep Onset (WASO) refer to the total number of minutes awake after first going to sleep and before waking up for the next day in the morning. Lower WASO corresponds to a better outcome.
  This endpoint measures the mean change from Weeks 1-2 to Weeks 9-10.
Mean Change in Total Sleep Time (TST) | 10 weeks
  Total sleep times (TST) refers to the total minutes of sleep starting at bedtime until waking up in the next morning. Higher TST corresponds to a better outcome.
  This endpoint measures the mean change from Weeks 1-2 to Weeks 9-10.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D Charlesworth, PhD, Study Director — Noctrix Health, Inc.
Locations (1):
- Noctrix Health Headquarters, Pleasanton, California, United States

IPD SHARING:
Plan to Share IPD: No
Due to the investigational nature of the device, IPD will not be shared for this study.